CLINICAL TRIAL: NCT00949000
Title: Clinical Evaluation of ST Segment Deviation Detection by SJM AnalyST and Analyst Accel Implantable Cardiac Defibrillators
Brief Title: AnalyST Treadmill Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Prof. Dr. Christian Hamm, Kerckhoff-Klinik
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CR08018HV
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ICD Implant (Other): Implantation of a commercially available AnalyST or AnalyST Accel ICD
  Interventions: Device: ICD Implantation

INTERVENTIONS:
Device: ICD Implantation — Implantation of a commercially available AnalyST or AnalyST Accel ICD

SUMMARY:
The objective of the study is to collect information on the naturally occurring variations in ST deviations at different heart rates, as detected by the AnalyST and AnalyST Accel Implantable Cardioverter Defibrillators (ICD).

ELIGIBILITY:
Inclusion Criteria:

* Patient has received or is scheduled to receive a St Jude Medical AnalyST or AnalyST Accel ICD;
* Patient has documented ischemic heart disease.

Exclusion Criteria:

* Patient has an indication for ventricular pacing;
* Patient has chronotropic incompetence or insufficiency;
* Patient has a contraindication to stress testing;
* Patient is physically unable to complete the stress test protocol;
* The patient has persistent or permanent atrial fibrillation (AF);
* Patient is unable to comply with the protocol and follow-up schedule based on geographic location or for any reason;
* Patient is pregnant;
* Patient is minor (< 18 years old).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of start and duration of isoelectric PR intervals | 4 weeks
Evaluation of start and duration of ST intervals | 4 weeks
Evaluation of ST segment deviations during stress testing across the 4 heart rate zones defined by the device | 4 weeks
Incidence of ischemic events detected based on the external ECG | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hamm, Prof. Dr., Principal Investigator — Kerckhoff-Klinik, Bad Nauheim, Germany
Locations (5):
- Germany (5):
  - Klinikum Coburg, Coburg, Bavaria
  - Kerckhoff-Klinik, Bad Nauheim, Hesse
  - Medizinische Einrichtungen der RWTH Aachen, Aachen, N. Rhin
  - Klinikum der Stadt Ludwigshafen am Rhein, Ludwigshafen, N. Rhin
  - Klinikum Luedenscheid, Lüdenscheid, N. Rhin